CLINICAL TRIAL: NCT02206581
Title: The Validity of Ultrasound Velocity to Detect Changes in the Hydration Status of Male and Female Athletes During Acute Dehydration and Rehydration
Brief Title: Using Hydration Monitor to Detect Changes in the Hydration Status Athletes
Status: Completed | Type: Observational
Sponsor: Artann Laboratories (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH); Appalachian State University (Other)
Responsible Party: Sponsor
Other Study IDs: HME-01; 2R44AG042990 (NIH)
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Dehydration
Keywords: dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- young healthy adult athletes: Hydration Monitor measurement of the ultrasound velocity and measures of hydration status including urine specific gravity, plasma and urine osmolality in male and female young adults after undergoing 3% acute dehydration and a 2-hr rehydration period
  Interventions: Device: Hydration Monitor

INTERVENTIONS:
Device: Hydration Monitor

SUMMARY:
The study will aim to evaluate the correlation between changes in ultrasound velocity and measures of hydration status including urine specific gravity, plasma and urine osmolality in male and female young adults after undergoing an acute dehydration and rehydration. The study will also test the hypothesis that body dehydration is a generalized physiological process equally affected all body muscles by comparing the data obtained on calf and biceps muscles.

ELIGIBILITY:
Inclusion Criteria:

* male or female athletes
* ages 18-25 years old

Exclusion Criteria:

* open wounds or rashes on calf testing area
* active skin infection
* pregnant female subjects

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The subject pool will be comprised of 100 young, healthy, physically active male and female subjects.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To observe statistically significant changes in ultrasound velocity associated with acute dehydration | 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Appalachian State University, Boone, North Carolina, United States